CLINICAL TRIAL: NCT07062380
Title: Prospective Validation of Multimodal Deep Learning Models for Predicting Recurrence Patterns in Early-Stage Hepatocellular Carcinoma After Resection: A Natural Treatment Cohort Stratification Study
Brief Title: AI-Based Prediction of HCC Recurrence Patterns After Resection (APAR)
Status: Recruiting | Type: Observational
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Wan-Guang Zhang, professor, Tongji Hospital
Other Study IDs: TJ-IRB202505060
Record Dates: First submitted 2025-07-02; First posted 2025-07-14 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-06

CONDITIONS: Hepatecellular Carcinoma; Hepatectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Surgery-Only Validation Cohort: Patients with early-stage HCC (BCLC 0-A) receiving curative liver resection without neoadjuvant/adjuvant therapy . Preoperative MRI, clinical data and pathological data will be used for AI model prediction of recurrence risk. Standard follow-up imaging for 2 years will validate model accuracy.
  Interventions: Procedure: Curative liver resection
- Exploratory Treatment Cohort: Patients with early-stage HCC receiving real-world neoadjuvant/adjuvant therapies (per physician discretion) alongside surgery. Treatment regimens and outcomes (RFS/OS) will be analyzed to assess therapy efficacy in model-stratified high/low-risk subgroups.
  Interventions: Procedure: Real-world multimodal therapy

INTERVENTIONS:
Procedure: Curative liver resection — Standard radical hepatectomy performed according to 2024 HCC guidelines. No neoadjuvant or adjuvant therapies administered. Follows institutional surgical protocols for BCLC 0-A HCC.
  Groups: Surgery-Only Validation Cohort
Procedure: Real-world multimodal therapy — Curative resection combined with clinically indicated therapies (e.g., TACE, targeted drugs, immunotherapy) as per treating physician's decision. Treatments recorded but not protocol-mandated.
  Groups: Exploratory Treatment Cohort

SUMMARY:
This observational study aims to validate a deep learning model for predicting aggressive recurrence patterns in patients with early-stage liver cancer (HCC) after surgery.

The main question it aims to answer is: Can the AI model accurately identify patients at high risk of cancer recurrence within 2 years after surgery? Participants will provide clinical data and undergo standard surgery, followed by 2-year imaging surveillance. Their data will be used for both AI prediction and validation of recurrence patterns.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-75 years, regardless of gender.
* BCLC stage 0-A, scheduled for curative liver resection.
* Preoperative clinical diagnosis of hepatocellular carcinoma (HCC).
* Availability of dynamic contrast-enhanced MRI within 1 month before surgery, with acceptable image quality.
* Child-Pugh liver function score ≤7.
* ECOG Performance Status (PS) 0-1.
* No severe organic diseases of the heart, lungs, brain, or other vital organs.

Exclusion Criteria:

* Concurrent other malignancies (except cured non-melanoma skin cancer or cervical carcinoma in situ).
* Postoperative pathology confirms non-HCC diagnosis.
* Pregnant or lactating women.
* History of organ transplantation.
* Inability to comply with the study protocol or follow-up schedule.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will enroll patients with early-stage hepatocellular carcinoma (BCLC 0-A) scheduled for curative liver resection at tertiary academic medical centers in China. Participants will be consecutively recruited from hepatobiliary surgery clinics, with preoperative MRI and postoperative pathology confirmation of HCC. The population reflects real-world clinical practice, including both surgery-only patients and those receiving neoadjuvant/adjuvant therapies per physician discretion.
Sampling Method: Non-Probability Sample
Enrollment: 353 (Estimated)
Dates: Start 2025-06-10 (Actual); Primary Completion 2026-06-10 (Estimated); Study Completion 2028-06-10 (Estimated)

PRIMARY OUTCOMES:
Accuracy of AI Model in Predicting Aggressive HCC Recurrence (AUC) | 2 years post-surgery
  The area under the receiver operating characteristic curve (AUC) of the multimodal deep learning model (PRE/POST) for predicting postoperative recurrence beyond Milan criteria within 2 years after resection, validated against actual imaging/histopathology-confirmed recurrence patterns.
  Unit : Dimensionless (0-1)

SECONDARY OUTCOMES:
Recurrence-Free Survival (RFS) | Up to 3 years
  Time from surgery to first radiologically confirmed recurrence (any pattern) or death from any cause, analyzed by Kaplan-Meier method and compared between model-predicted high/low-risk groups.
  Unit : Months
Overall Survival (OS) | Up to 5 years
  Time from surgery to death from any cause, compared between patients stratified by AI model predictions (high-risk vs. low-risk) and treatment cohorts (surgery-only vs. real-world therapy).
  Unit : Months

OTHER OUTCOMES:
Therapeutic Efficacy in Exploratory Cohort | Up to 1 years
  Objective response rate (ORR) and RFS/OS benefits of neoadjuvantin model-predicted high-risk patients, assessed descriptively (non-randomized comparison).
  Unit : Percentage (%)

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji Hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No